CLINICAL TRIAL: NCT01706848
Title: A Post Market Clinical Study Evaluating the Safety, Device Performance and Possible Emergent Risks of Celotres in the Improvement of Wound Healing and the Resulting Scar Consequences Following Suturing of a Wound
Brief Title: Celotres for Improvement in Wound Healing and Resulting Scar Consequences Following Suturing of a Wound
Acronym: PMCS EURO HEAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Halscion, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HAL-0297
Record Dates: First submitted 2012-10-03; First posted 2012-10-15 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2013-08

CONDITIONS: Scar
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Celotres (Active Comparator): Scar halves randomized to treatment with device, opposite side treated per standard of care.
  Interventions: Other: Celotres
- Standard surgical wound closure (Active Comparator): Scar halves randomized to treatment with device, opposite side treated per standard of care.
  Interventions: Other: Surgical Closure by Standard of Care

INTERVENTIONS:
Other: Celotres — Surgical procedure will be performed as per the standard of care. Scar halves randomized to treatment with device (Celotres), opposite side treated per standard of care.
  Arms: Celotres
Other: Surgical Closure by Standard of Care — Surgical procedure will be performed as per the standard of care. Scar halves randomized to treatment with device (Celotres), opposite side treated per standard of care.
  Arms: Standard surgical wound closure

SUMMARY:
The objective of the study is to actively gather additional information on safety, device performance and possible emergent risks following the use of Celotres in a post-market setting when used to improve wound healing and the resulting scar consequences following suturing of a wound.

ELIGIBILITY:
Inclusion Criteria:

* Patients electing to undergo a surgical procedure;
* Patients able and willing to give written informed consent

Exclusion Criteria:

* Patients with a known or potential risk of allergy or sensitivity to products or substances containing porcine gelatin

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-09; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Safety | Assessed at treatment, suture removal, Months 1, 3, 6, 9 and 12
  Safety as defined by the incidence of device related adverse events.

SECONDARY OUTCOMES:
Effectiveness | Assessed at Months 1, 3, 6, 9 and 12
  Patient and Observer Scar Assessment Scale (POSAS)
Device Performance Evaluation | Assessed at Day 1
  Questions related to packaging integrity and successful administration of product as assessed by the Principal Investigator

CONTACTS AND LOCATIONS:
Overall Officials: Venkat Ramakrishnan, MD, Principal Investigator — Brentwood Hospital
Locations (9):
- Poland (3):
  - Angelius Szpital Proviat, Katowice
  - Oddzial Leczenia Oparzen Chirugil Plastysznej, Krakow
  - Wojskowy Oddzial Kliniczny ChirurgiiPlastycznej, Warsaw
- United Kingdom (6):
  - The Westbourne Center, Birmingham
  - Brentwood Hospital, Brentwood
  - Plastic Surgery W1 Ltd, Suite 1, London
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - Norfolk and Norwich University Hospital, Norwich
  - Morriston Hospital, Swansea